CLINICAL TRIAL: NCT03518112
Title: Phase II Study of the Combination of Low-Intensity Chemotherapy and Blinatumomab in Patients With Philadelphia Chromosome Negative Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Low-Intensity Chemotherapy and Blinatumomab in Treating Patients With Philadelphia Chromosome Negative Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Competing Studies
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0127; NCI-2018-00737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0127 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Philadelphia Chromosome Negative; Recurrent B Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegfilgrastim; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (blinatumomab, combination chemotherapy) (Experimental): See detailed description.
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Biological: Pegfilgrastim; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; BW 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well low-intensity chemotherapy and blinatumomab work in treating patients with Philadelphia chromosome negative acute lymphoblastic leukemia that has come back or does not respond to treatment. Drugs used in chemotherapy, such as dexamethasone, filgrastim, pegfilgrastim, cyclophosphamide, methotrexate, cytarabine and vincristine sulfate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as blinatumomab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving low-intensity chemotherapy and blinatumomab may work better at treating acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the combined effect of blinatumomab and mini-hyper-CVD (low-intensity chemotherapy) on event-free survival.

SECONDARY OBJECTIVES:

I. Evaluating other clinical efficacy endpoints (minimal residual disease [MRD] negativity, duration of response, the overall response rate [complete response (CR) + CR with inadequate count recovery (CRi)]) of the regimen occurred any time during the treatment.

II. Overall survival. III. Determining the safety of the combination regimen.

OUTLINE:

INDUCTION PHASE: Patients receive blinatumomab intravenously (IV) continuously on days 1-28 and dexamethasone orally (PO) or IV over 30 minutes on days -3 to day 0 and 7-10. Patients also receive filgrastim subcutaneously (SC) on days 1-42 or pegfilgrastim SC on days 1 and 25, cyclophosphamide IV over 3 hours twice daily (BID) on days -3 to -1, methotrexate intrathecally (IT) on day 2 and IV over 24 hours on day 22, cytarabine IT on day 7 and IV over 3 hours BID on days 23 and 24, and vincristine sulfate IV over 15 minutes on days 0 and 7. At the discretion of the treating physician, patients may receive rituximab IV over 4-6 hours on days -3, 0, 22 and 29, and leucovorin calcium IV over 15 minutes or PO 4 times daily (QID) for 8 doses.

CONSOLIDATION PHASE: Patients receive blinatumomab IV continuously on days 1-28 and dexamethasone PO or IV over 30 minutes on days 1-4 and 11-14. Patients also receive cyclophosphamide IV over 3 hours BID on days 1-3, vincristine sulfate IV over 15 minutes on days 1 and 11, filgrastim SC on days 1-4 and 22-42 or pegfilgrastim SC on day 5 and 25, methotrexate IT on day 2 and IV over 24 hours on day 22, cytarabine IT on day 7 and IV over 3 hours BID on days 23 and 24. At the discretion of the treating physician, patients may receive rituximab IV over 4-6 hours on days 1, 8, 22 and 29, and leucovorin calcium IV over 15 minutes or PO QID for 8 doses. Treatment repeats every 42 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive prednisone PO and vincristine sulfate IV over 15 minutes on days 1-5 of cycles 5-9, 7-11 and 13-24, and mercaptopurine PO BID on days 1-28 of cycles 1-5, 7-11, and 13-24. Patients also receive methotrexate PO once a week and blinatumomab IV continuously on days 1-28 of cycles 6 and 12. Cycles repeat every 28 days for up to 24 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first or second relapsed/refractory B-cell acute lymphoblastic leukemia (ALL)
* Performance status =< 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the principal investigator (PI)
* Alanine aminotransferase (ALT) =< 3 x ULN, unless due to the underlying leukemia approved by the PI
* Aspartate aminotransferase (AST) =< 3 x ULN unless due to the underlying leukemia approved by the PI
* Signed informed consent
* Women of childbearing potential (WOCBP) or male subjects with a partner who is WOCBP must agree to use contraception during the study, if sexually active

Exclusion Criteria:

* Patients with Philadelphia chromosome (Ph)-positive ALL or Burkitt leukemia
* Active, uncontrolled central nervous system (CNS) leukemia involvement
* Active serious infection not controlled by oral or intravenous antibiotics
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Known hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Patients with a cardiac ejection fraction (as measured by either multi-gated acquisition [MUGA] or echocardiogram) < 40%
* Prior history of treatment with blinatumomab
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last two weeks, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception; women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months; in addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2018 to May 2021
Period: Overall Study
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 47 [33 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS) Where Events Defined as no Response, Loss of Response, or Death
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse. Relapse and resistant disease will be defined based on morphological assessment of bone marrow and peripheral blood.
  Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR.
  Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
  Partial Response (PR): As above for CR except for the presence of 6-25% marrow blasts.
Time Frame: Time from the first day of treatment assessed up to 3 years, 1 month
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 5
Months | 5.7 [1.4 to 34.7]

2. Secondary Outcome: Number of Participants Negative for Minimal Residual Disease (MRD)
Description: Minimal Residual Disease (MRD) was assessed by flow cytometry. MRD negativity: Absence of detectable leukemia using multiparameter flow cytometry with a sensitivity of </= 0.01%.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Duration of Response
Description: Response date to loss of response or last follow up. Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR.
  Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
  Partial Response (PR): As above for CR except for the presence of 6-25% marrow blasts.
Time Frame: Time from the first day of treatment assessed up to 3 years, 1 month
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 4
Months | 4.4 [1.2 to 34.7]

4. Secondary Outcome: Participants With a Response
Description: defined as the percentage of patients achieving complete response (CR) or CR with inadequate count recovery (CRi). Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR.
  Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 5
Participants | 4

5. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Time from the first day of treatment assessed up to 3 years, 1 month
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
Number analyzed (Participants) | 5
Months | 16.7 [6.9 to 37]

ADVERSE EVENTS:
Time Frame: Time from the first day of treatment assessed up to 3 years, 1 month
Arm/Group | Treatment (Blinatumomab, Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Blinatumomab, Combination Chemotherapy) (N=6)
Fever (General disorders) | 2 (3)
Headache (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Concentration Impairment (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Night Sweats (General disorders) | 1 (1)
Edema Legs (General disorders) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (2)
Thrombocytopenia (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Neutopenia (Blood and lymphatic system disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased White Blood Count (Blood and lymphatic system disorders) | 2 (3)
Cytokine Release Syndrome (Immune system disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Steroid Myopathy (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03518112/Prot_SAP_000.pdf